CLINICAL TRIAL: NCT06624397
Title: Evaluation of a Skills-Based Program for Carers & Families of Patients with Anorexia Nervosa
Brief Title: Evaluation of a New Program for Carers of People with Anorexia Nervosa
Acronym: CAREFREE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Forth Valley (Other Government)
Collaborators: NHS Lothian (Other Government); University of Stirling (Other); NHS Greater Glasgow and Clyde Board HQ (Other)
Responsible Party: Principal Investigator, Dr Susan Simpson, Consultant Clinical Psychologist, NHS Forth Valley
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: FV1421; TCS/22/05 (Other Grant/Funding Number: Chief Scientist Office, Scottish Government)
Record Dates: First submitted 2024-09-23; First posted 2024-10-03 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-09

CONDITIONS: Anorexia Nervosa; Carer Stress Syndrome
Keywords: Anorexia Nervosa; Burnout; Carer Burnout; CAREFREE
MeSH Terms: conditions — Anorexia Nervosa; Burnout, Psychological

STUDY DESIGN:
Intervention Model Description: CAREFREE is a 12-session Carer's Programme for carers of adults with moderate to severe Anorexia Nervosa. This programme was developed to provide carers with an opportunity to develop an understanding of Anorexia from a Biopsychosocial framework, taking into account the complex array of biological, psychological and social/environmental factors associated with the development and maintenance of this disorder. CAREFREE is based on a Schema Therapy - Compassion Focused framework, incorporating psychoeducation in regard to both Anorexia Nervosa and Carer Burnout. The programme has a relational focus, with an emphasis on improving emotional fluency, family communication skills and self-other compassion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CAREFREE is a 12-session Carer's Programme (Experimental): This programme was developed to provide carers with an opportunity to develop an understanding of Anorexia from a Biopsychosocial framework, taking into account the complex array of biological, psychological and social/environmental factors associated with the development and maintenance of this disorder. CAREFREE programme is unique in its focus on providing a framework for understanding AN from a Schema Therapy - Compassion Focused framework, incorporating psychoeducation in regard to both Anorexia Nervosa and Carer Burnout. The programme has a relational focus, with an emphasis on improving emotional fluency, family communication skills and self-other compassion.
  Interventions: Other: CAREFREE Carer's Programme

INTERVENTIONS:
Other: CAREFREE Carer's Programme — This programme was developed to provide carers with an opportunity to develop an understanding of Anorexia from a Biopsychosocial framework, taking into account the complex array of biological, psychological and social/environmental factors associated with the development and maintenance of this disorder. CAREFREE programme is unique in its focus on providing a framework for understanding AN from a Schema - Compassion Focused framework, incorporating psychoeducation in regard to both Anorexia Nervosa and Carer Burnout. The programme has a relational focus, with an emphasis on improving emotional fluency, family communication skills and self-other compassion.

SUMMARY:
CAREFREE is a 12-session Carer's Programme for carers of adults with moderate to severe Anorexia Nervosa. This programme was developed to provide carers with an opportunity to develop an understanding of Anorexia from a Biopsychosocial framework, taking into account the complex array of biological, psychological and social/environmental factors associated with the development and maintenance of this disorder. The CAREFREE programme is unique in its focus on providing a framework for understanding AN from a Schema -Compassion Focused framework, incorporating psychoeducation in regard to both Anorexia Nervosa and Carer Burnout. The programme has a relational focus, with an emphasis on improving emotional fluency, family communication skills and self-other compassion. The CAREFREE programme is open to carers from across Scotland and runs online. Outcomes (including carer and patient quality of life, family communication, patient motivation to change) will be analysed and published at the end of the 24-month period. One of the key benefits of this programme is that as it is a cross-regional-NHS project.

DETAILED DESCRIPTION:
Moderate to Severe Anorexia Nervosa (AN-MS)is characterised by poor treatment outcomes, poor quality of life, low motivation levels and ambivalence about change, with high burden on families and NHS services. This study aims to improve quality of life and relationships amongst those with AN-MS and their families/partners/carers, and enhance motivation to recover amongst adults with AN-MS, ultimately resulting in enhanced care and reduced inpatient admissions. We will evaluate a new online group intervention for families/carers and partners. This is a two-phase study: Phase 1 feasibility trial will evaluate factors such as recruitment and retention of clinicians and participants, collection of assessment measures and acceptability of the intervention. Phase 2 will use this information to inform the development of a second more robust feasibility study which will enable us to determine whether this new untested intervention is effective in its own right, as a precursor for a larger definitive trial.

ELIGIBILITY:
Carer Participants

Inclusion Criteria

* Has a family member, partner or spouse/partner with moderate-severe, treatment resistant and/or co-morbid anorexia nervosa (as diagnosed by a clinician at one these centres)
* Is over the age of 17
* Can speak and read English
* Has access to the internet and is comfortable using an online meeting platform

Exclusion Criteria

* Cannot speak/read English
* Is currently suffering from acute psychosis

Participants with Anorexia

Inclusion Criteria

* Have moderate-severe, treatment resistant and/or co-morbid anorexia nervosa (as diagnosed by a clinician at one these centres)
* Is over 17 years of age
* Can speak and read English

Exclusion Criteria

• Is currently suffering from acute psychotic mental health state

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
(SRS-Version 3) (Johnson, Miller, & Duncan, 2000). | Weekly after each Carer group Session
  Therapeutic alliance will be evaluated using this 4-item Session Rating Scale after each session
Short Rating Scales | Pre (0-6 weeks before group programme begins); Weekly throughout programme; and Post (0-4 weeks after group programme ends)
  - VAS scales will used to assess carers' ratings of: (1) Quality of life (taken from the WHOQOL-BREF) and (2) Quality of relationship with the patient with AN. (taken from SCORE-15)
Experiences in Close Relationships Revised (ECR-R; Fraley et al., 2000; 36 items) | Pre (0-6 weeks before group programme begins) and Post (0-4 weeks after group programme ends) and at 3-months followup
  Assesses self reported individual differences regarding attachment-related anxiety and avoidance.
WHOQOL-BREF (WhoQol Group, 1998) | Pre (0-6 weeks before group programme begins); Post (0-4 weeks after group programme ends) and at 3-months followup
  This is a World Health Organisation Quality of Life Assessment and is a widely used quality of life instrument which contains 26 items over 4 dimensions - physical health, psychological health, social relationships, environment, quality of life and general health.
Depression, anxiety, and stress scale (DASS) | Pre (0-6 weeks before group programme begins); Post (0-4 weeks after group programme ends) and at 3-months followup
  Depression, anxiety, and stress scale (DASS) is a 21-item measure assessing depression, anxiety, and stress over the past seven days using a four-point Likert scale. Scores of these three subscales can be added to obtain a total score for psychological distress.
SCORE-15 Index of Family Functioning and Change (Stratton et al., 2010) | Pre (0-6 weeks before group programme begins); Post (0-4 weeks after group programme ends) and at 3-months followup
  - SCORE is a self report outcome measure designed to be sensitive to the kinds of changes in family relationships that systemic family and couples' therapists see as indications of useful therapeutic change.
Family Questionnaire (Wiedemann et al 2002) | Pre (0-6 weeks before group programme begins); Post (0-4 weeks after group programme ends) and at 3-months followup
  This questionnaire will be used to measure expressed emotion within the family system.
Schema Mode Inventory (Young et al., 2007) | Pre (0-6 weeks before group programme begins); Post (0-4 weeks after group programme ends) and at 3-months followup
  5 items of this scale are included in the outcomes to measure healthy functioning.
Eating disorder symptom impact scale (EDSIS; Sepulveda et al., 2008) | Pre (0-6 weeks before group programme begins); Post (0-4 weeks after group programme ends) and at 3-months followup
  This is a 24-item self-report measure of caregiving burden in eating disorders. The scale comprises of subjective and objective burden across four subscales: managing nutritional situations, dealing with dysregulated behaviors, guilt, and social isolation. Scores are obtained on a five-point Likert scale. Higher scores indicate higher caregiving burden and more negative appraisal of caregiving
Young Parenting Inventory-revised (YPI-R2; Louis, Wood and Lockwood, 2018) | Pre -group (0-6 weeks before group programme begins)
  This scale assesses perceived parenting experiences. The YPI-R2 is a 36-item questionnaire measuring parenting styles, namely: Competitiveness and Status seeking; Degradation and Rejection; Emotional Inhibition and Deprivation; Overprotection and Overindulgence; Punitiveness; Controlling. Subscale scores are calculated as mean scores with higher scores indicating stronger perceived negative parenting.

SECONDARY OUTCOMES:
Eating Disorder Quality of Life questionnaire (EDQoL; Engel et al., 2006). | Pre (0-6 weeks before group programme begins) and Post (0-4 weeks after group programme ends)
  Measures Quality of Life of the Patient with Anorexia Nervosa
SCORE-15 and Young Parenting Inventory (YPI-R)) | Pre (0-6 weeks before group programme begins); and Post (0-4 weeks after group programme ends)
  These measure family functioning in the patient with Anorexia Nervosa
Anorexia Nervosa Stages of Change Questionnaire (ANSOCQ; Rieger et al., 2002) | Pre (0-6 weeks before group programme begins); and Post (0-4 weeks after group programme ends)
  This scale measures motivation to recover in the person with Anorexia Nervosa
Demographics Questionnaire | 0-6 weeks before attending group programme
  A demographics questionnaire will be filled out by the person with Anorexia Nervosa to ascertain details including: age, age of onset of eating disorder, occupation, relationship with the patient/carer, level of education, postcode, whether or not the person with anorexia is living from home and/or what age they moved out; relationship status, receipt of patient/carer benefits.
Qualitative Interview with person with Anorexia Nervosa | 0-4 weeks after group intervention is completed
  A Qualitative Interview will be carried out with the person with Anorexia Nervosa whose carers are attending the CAREFREE programme, to ascertain their views on the degree to which the programme has impacted family functioning and relationships, as well as their own perspectives in regard to Anorexia Nervosa.

OTHER OUTCOMES:
Carer Qualitative interviews and Focus Groups | Focus groups will be carried out immediately following Sessions 6 and 12 - 6 weeks and 12 weeks into the intervention.
  Focus groups will focus on quality of life and the achievement of personalised treatment goals (developed with group leaders) will be conducted with carer participants at Mid- and Post- Intervention
Feasibility observations | Feasibility measures will be evaluated immediately following the completion of the Group Programme (i.e. following Session 12 at week 12 of the programme).
  - What is the feasibility (uptake, retention, dropout, acceptability) of running a novel 12-week group programme for carers, partners and family members of individuals with moderate-severe, treatment resistant and co-morbid AN?(a) Can the investigators recruit clinicians to take part in the study? Can the investigators implement study procedures correctly? Can the investigators implement the intervention with adequate fidelity? (b) Can the investigators recruit patients to the study? How many participants are excluded by the eligibility criteria? How many participants drop out before the end of the study? Can participants complete the assessments? Do participants comply with the intervention? How much missing data is there? (c) What estimates of effect size/variability should be used in the design of the full study?(d) According to carer participant perspectives, what are the most useful aspects of the programme?

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - NHS Glasgow, Glasgow, Scotland
  - NHS Forth Valley, Stirling, Stirlingshire

IPD SHARING:
Plan to Share IPD: Undecided
De-identified patient data will only be shared with researchers who are directly involved in the project in some capacity